CLINICAL TRIAL: NCT03276689
Title: 'Fix the Dysfunction' Concept for Mechanism-based Pharmacological Treatment of Neuropathic Pain by Drug
Acronym: 0381-16
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Israel Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0381-16-RMB_CTIL
Record Dates: First submitted 2017-08-30; First posted 2017-09-08 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Treatments The patients will take 2 tab/d of either (i) duloxetine 60mg or (ii) pregabaline 150mg x 2/day or (iii) placebo for 8 weeks. In the first 7 days dose of duloxetine will be 30mg/day in order to lower side effects and improve compliance. In line, the initial 7-days dose of pregabaline will 75mg x 2. For duloxetine, the morning dose will be a sham pill. Study nurse will be available for the patients regarding any side effects or issues arising, and communicate the relevant data to the PI. All personnel and patients will be blinded to the given treatment (double-blind design). The person conducting the immediate and the long term follow up will not know what the results were of the pre-treatment assessments.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All personnel and patients will be blinded to the given treatment (double-blind design). The person conducting the immediate and the long term follow up will not know what the results were of the pre-treatment assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Duloxetine (Experimental): The patients will take 2 tab/d of duloxetine 60mg for 8 weeks. In the first 7 days dose of duloxetine will be 30mg/day in order to lower side effects and improve compliance. For duloxetine, the morning dose will be a sham pill.
  Interventions: Drug: Duloxetine
- Pregabaline (Experimental): The patients will take 2 tab/d of pregabaline 150mg x 2/day for 8 weeks.The initial 7-days dose of pregabaline will 75mg x 2.
  Interventions: Drug: Pregabaline
- Placebo (Experimental): The patients will take 2 tab/d placebo for 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Duloxetine — The patients will take duloxetine for 8 weeks.
  Arms: Duloxetine
Drug: Pregabaline — The patients will take pregabaline for 8 weeks.
  Arms: Pregabaline
Other: Placebo — The patients will take placebo for 8 weeks.
  Arms: Placebo

SUMMARY:
Introduction Treatment of neuropathic pain has been a goal of numerous research projects for the last half century, with overall disappointing results. These poor achievements are in contrast with substantial advancements in the understanding of pain mechanisms, and numerous molecules developed to tackle them. The need to better identify patients likely to respond to treatment comes from the neuropathic pain experts in regards to the pharmacological domain.

The basic assertion of this project is that the pain modulation profile is altered in pain patients toward a pro-nociceptive mode, and that the specific single or multiple dysfunctions of pain modulation that underlie this pro-nociceptivity should be targeted by therapeutic lines that can reverse the modulation back toward eu-nociceptivity.

The aim of this amendment is to demonstrate that pain treatment efficacy for painful diabetic neuropathy can be optimized by individualizing pharmacological treatment choice along 'fix the dysfunction' concept

DETAILED DESCRIPTION:
Introduction Treatment of neuropathic pain has been a goal of numerous research projects for the last half century, with overall disappointing results. These poor achievements are in contrast with substantial advancements in the understanding of pain mechanisms, and numerous molecules developed to tackle them. The need to better identify patients likely to respond to treatment comes from the neuropathic pain experts in regards to the pharmacological domain.

The basic assertion of this project is that the pain modulation profile is altered in pain patients toward a pro-nociceptive mode, and that the specific single or multiple dysfunctions of pain modulation that underlie this pro-nociceptivity should be targeted by therapeutic lines that can reverse the modulation back toward eu-nociceptivity.

The aim of this amendment is to demonstrate that pain treatment efficacy for painful diabetic neuropathy can be optimized by individualizing pharmacological treatment choice along 'fix the dysfunction' concept Methods Study design This is a longitudinal double blind non cross over study with parallel groups. There will be three pharmacological treatment arms, one per each treatment: SNRIs duloxetine, Ca++-channels blocker pregabaline and inactive placebo. All treatments will be given to painful diabetic neuropathy patients. All patients will undergo three lab sessions. A uniform assessment will be performed before starting (Session I), and at the end of treatments (Session III). This psychophysical assessment of their pain modulation, physiological assessment that will include resting-state EEG recording along with contact-heat evoked potentials (CHEPs) and assessment of motor cortex excitability, and psychological assessment with pain-related psychological questionnaires. In addition, Session I will also include a clinical examination for the assessment of neuropathy characteristics and symptoms severity.

After one months after the initial Session I, all the patients will undergo the lab session for the assessment their responsiveness to experimental placebo manipulation (Session II), including filling questioners associated with the prediction of placebo effect.

Between sessions I and II the patients will fill an electronic diary in order to evaluate their clinical pain intensity.

A group of age- matched healthy subjects will undergo a psychophysical pain modulation protocol along with the EEG recording, all performed in one session. These data will serve a reference data for this study.

Patients Three-hundred Painful Diabetic Neuropathy patients will be recruited. Inclusion criteria: age of 18-80 yrs, both genders, non-pregnant or breast feeding, free of significant chronic pain syndromes other than the neuropathy, free of major neurological or psychiatric disorders such as dementia, psychosis and similar. Exclusion criteria: communication and language difficulties that hinder their performance in the various tests.

One-hundred healthy subjects will be recruited. Inclusion criteria: age of 18-80 yrs, both genders, non-pregnant or breast feeding, free of significant chronic pain syndromes, free of major neurological or psychiatric disorders such as dementia, psychosis and similar. Exclusion criteria: communication and language difficulties that hinder their performance in the various tests.

Assessment of neuropathy and baseline pain Clinical evaluation will be based on a clinical interview and examination, data will be collected using the Toronto scale. Assessment of pain along four weeks will be recorded via a smart phone application on weekly basis, , or by follow up phone calls to patients/ printed diary. Quantitative sensory testing (thermal sensory thresholds assessment) and/or EMG assessment will be performed on the most affected foot in order to evaluate neuropathy severity. QST-wise we will follow the DFNS for the following items: Sensory and pain thresholds. tested with 3x3cm contact Peltier probe of the Thermal Sensory Analyzer (TSA, Medoc, Israel) device. The baseline temperature will be set at 32oC; with stimulus change rate of 1 oC/sec for the assessment of sensory and pain threshold. Thresholds for heat and cold pain will be measured using method of limits, based on the mean of 3 responses. Mechanical sensory and pain threshold will be assessed with von Frey filaments (Bioseb, France) applied in an ascending order at several repetitions. Five threshold determinations will be made, each with a series of ascending and descending stimulus intensities. The final threshold is the geometric mean of these five series of supra- and subthreshold stimuli intensities. Dynamic mechanical allodynia using standard brush. Vibration detection threshold (VDT). This test is performed with a standardized tuning fork (64 Hz) that is placed on the toes and patella. The vibration detection threshold is determined by three series of descending stimulus intensities determined from the "wandering" tip of a triangle moved by means of the vibration and indicated on the tuning fork using the arithmetic mean of the values when the participant just stopped perceiving vibration (in x/8). Pressure pain threshold (PPT). Using a pressure algometer (contact area 1 cm2) the threshold for pressure induced pain is measured above a foot muscle in 3 series of slowly increasing stimulus intensities (0.5 kg/s, corresponding to 50 kPa/s). The threshold is then determined as the arithmetic mean of the 3 series (in kPa).

Psychophysical pain modulation protocols CPM response will be assessed by two test-stimuli: (i) contact heat, a 10" contact heat stimulus (30x30 mm thermode, TSA-2001, Medoc, Israel) delivered to the left forearm at the individually-predetermined temperature that evoked pain intensity of 60 on a 0-100 NPS. (ii) mechanical stimuli, three application of pressure algometer device, Algomed, Medoc Israel), for 1" each delivered with the inter-stimulus interval (ISI) of 5" (to prevent summation). Conditioning stimulus will be cold water immersion of the other hand in a water container of 8-10oC. Alternatively, the test- and conditioning stimuli might be applied on upper or/and lower back. In addition, instead of cold water we might use a contact heat stimuli or ice package. After short familiarization with the various stimuli, each test-stimulus will be administered, and response measured. A 10' break will be taken, and then the conditioning stimulus will be given, during which the three test stimuli will be repeated. The difference between conditioned test stimulus result and the stand alone result will be the taken as the CPM effect. Please see https://www.youtube.com/watch?v=jL9GgdsyHtA for our detailed protocol.

TS response will be measured on the left forearm using two tests: (i) mechanical stimuli; application of a 180gr (# 6.45) von Frey filament. NPS will be obtained after a single application, and after the last application in the series of 10 repetitive stimuli with a 1" inter-stimulus interval. (ii) electrical stimuli, a series of a single, and then of 10 electrical stimuli will be given at the intensity of Pain50 and ISI of 1", using the stimulation parameters as described for NFR (iii) tonic heat stimulus of 50/100 for 30" with ratings along the stimulus. The difference between the last and the first scores for each type of stimulus will be taken as the TS score. In addition, magnitude estimation of supra-threshold pain with tonic stimuli of 45oC, 47oC and 49oC, 10" each, and pain scores in response to hand immersion will serve as the static pain parameters of pain sensitivity.

EEG protocol Resting-state EEG and contact heat-evoked potentials (CHEPs) will be recorded with 64 channels ActiChamp EEG system (Brain Products GmbH, Munich, Germany). The data will be saved on hard disk for offline analysis.

CHEPs will be recorded for all of the following 'test stimuli'. These will be phasic stimuli (PATHWAY system, Medoc, Israel), delivered to the forearm, rising at 70oC/sec with immediate return to adaptation, with peak intensity at predetermined temperature evoking pain60. For the neurophysiological assessment of CPM, there will be two blocks of stimuli; each consisting of 30 stimuli, divided into two trains of 15 stimuli separated by 5', ISI is 8-12". Pain ratings will be obtained in parallel to the recording of CHEPs, after each stimulus. The first block will be given as a stand-alone; the second one will be given in parallel to immersion of the other hand in cold water of 8-10oC as the 'conditioning stimulus'. Alternatively, a tonic contact heat or ice package application will serve a conditioning stimulus. The CPM effect will be the difference between the current density maps of the CHEPs in response to test-stimuli given before and during conditioning-stimuli. EEG analysis: Source localization of brain generators will be pursued by sLORETA (free academic software at: http://www.uzh.ch/keyinst/loreta.htm) to compute statistical non-parametric maps from the contact heat and electrical pain evoked potentials aimed to identify the most active cortical areas related to the CPM. After identifying the regions of interest (ROI's) based on their putative role in pain inhibitory and facilitatory modulation processing, S-LORETA will calculate the average current density value for the ROI or the voxel with maximal activity for each patient, based on the individual electrode coordinates.

EEG frequency analysis. Each 3-minute resting-state recording section will be divided into segments of 1 second. Segments contaminated with eye movements, muscle activity or other artifacts will be removed from further analysis. The remaining segments will be subject to time frequency analysis using wavelet transform i.e. decomposition of the signal to different wavelet templates each represent a combined time-frequency representation and each assigned a coefficient according to its match with the original signal. We will use the coefficients (averaged over time) to calculate the frequency content power and peak frequency for each of the following frequency bands: delta (2-4Hz), theta (4-8Hz), alpha 1 (8-10Hz), alpha 2 (10-12Hz), beta (13-25Hz) and gamma (>30Hz). The coefficients of the signal at different scalp location can be used to calculate phase synchronization and the coherence of the activity between different brain regions reflecting functional connectivity among related brain regions.

Treatments The patients will take 2 tab/d of either (i) duloxetine 60mg or (ii) pregabaline 150mg x 2/day or (iii) placebo for 8 weeks. In the first 7 days dose of duloxetine will be 30mg/day in order to lower side effects and improve compliance. In line, the initial 7-days dose of pregabaline will 75mg x 2. For duloxetine, the morning dose will be a sham pill. Study nurse will be available for the patients regarding any side effects or issues arising, and communicate the relevant data to the PI. All personnel and patients will be blinded to the given treatment (double-blind design). The person conducting the immediate and the long term follow up will not know what the results were of the pre-treatment assessments.

Placebo-manipulation session During session II we will perform an evaluation of placebo responsiveness as follows. First, the patient will be exposed to moderate noxious individually-tailored heat stimulus (up to 1 min duration) given on the dominant forearm. After topical application of a neutral hand cream (like Vaseline), which will be presented to the participants in advance as a very powerful analgesic cream, 15 min break will be taken after which the subject will told that the cream will be active for next 30-40 min during which repeated assessment of pain perception will be performed. First, lower intensity of the heat stimulus will be given (a conditioning procedure). Then, with a further 10 min break, two stimuli of the initially chosen temperature will be delivered, and pain perception will be assessed. The placebo response will be calculated as a pain reduction between post- vs. pre-conditioning heat pain application. The participants also rate their expectation of the painfulness before, and the actually perceived pain after each heat stimulus.

During this session all patients will also undergo the psychological assessment as follows: Anxiety, pain-related catastrophizing and sleep quality will be assessed via the relevant questioners of the set of psychological assessment developed for our undergoing Horizon 2020 study. In addition, all participants will fill the Multidimensional Iowa Suggestibility Scale (MISS) questioner for the assessment of individual suggestibility.

In addition to the psychological evaluation, the patients will undergo cognitive / attentional assessment of cognitive flexibility and working memory using the Trail-Making Test A and B parts, and the Digit Symbol Submission Test.

Follow-up Longitudinal assessment of clinical pain level will be reported every two weeks along 8 weeks of the treatment, via a smart phone application that will be downloaded to participating patient's devices, or by follow up phone calls to patients/ printed diary . In addition - the full assessment lab protocol performed at baseline will be repeated at the end of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* age of 18-80 yrs,
* both genders, * non-pregnant or breast feeding,
* free of significant chronic pain syndromes other than the neuropathy,
* free of major neurological or psychiatric disorders such as dementia, psychosis and similar.

Exclusion Criteria:

*communication and language difficulties that hinder their performance in the various tests.

One-hundred healthy subjects will be recruited, with the same inclusion exclusion criteria.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Pain modulation | During 8 weeks of treatment, every 2 weeks and at the end of the treatment, meaning after 8 weeks from day 1 of the start of medication
  Pain will be measured by using VAS scale from 0 - 100. Resting-state EEG recording along with contact-heat evoked potentials (CHEPs) and assessment of motor cortex excitability, and psychological assessment with pain-related psychological questionnaires, will be collected. .

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No